CLINICAL TRIAL: NCT03486184
Title: Postoperative Acute Kidney Injury in Patients Undergoing Prolonged Neurosurgical Operations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Maher Abdel Salam Ahmed, Resident, Assiut University
Other Study IDs: acute kidney injury
Record Dates: First submitted 2018-03-22; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Postoperative Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cystatin-C — * Laboratory values will be obtained, including level of preoperative serum creatinine, complete blood count, coagulation profile and Cystatin-C (5 ml. venous sample).
  * Serum creatinine and hemoglobin will be measured after operation, and thereafter at least once a day as a part of routine clinical care. Postoperative serum Cystatin-C will measured only once.

SUMMARY:
Postoperative Acute Kidney Injury in Patients Undergoing Prolonged Neurosurgical Operations

DETAILED DESCRIPTION:
* Postoperative acute kidney injury (AKI) is a highly prevalent and prognostically important complication in various surgical settings. Patients who developed postoperative AKI is independently associated with markedly increased morbidity, mortality1-8 and higher economic burden1.
* AKI was defined by an increase in serum creatinine (SCr) ≥ 0.3 mg/dl or by an increase in SCr ≥ 50% and/or by a decrease in urine output to 0.5 ml/kg/hour for 6 hours, in the first 48 hours after surgery.
* Patients who developed AKI had a higher total ICU costs, prolonged length of hospital and ICU stay, and longer duration of postoperative mechanical ventilation.
* AKI has been studied in different surgical procedures especially cardiac & abdominal surgeries.
* Kovacheva et al 2016 retrospective study included 1656 craniotomy patients from 1998 to 2011. The AKI used criteria was RIFLE (Risk, Injury, Failure, Loss of kidney function and End-Stage Renal Failure), they reported an incidence of 9.9% of postoperative AKI9.
* Deng et al 2017 also reported an incidence of AKI up to 13.5% in patients undergoing neurosurgical surgery within the first 7 days. It was associated with independent risk factors included intraoperative blood loss, postoperative reoperation, use of mannitol during operation, concentration of Cystatin-C; a biomarker protein detecting early kidney injury before creatinine changes and postoperative APACHE II score10.
* As the number of neurosurgical procedures has been increased worldwide and in our department as well with new types of prolonged neurosurgery e.g. Skull - Base - Major cerebrovascular beside major cranial tumor excision. It becomes a necessary to re-evaluate the incidence, factors behind AKI and outcome in such prolonged surgery.
* In 2002, The Acute Dialysis Quality Initiative (ADQI) was created with primary goal was to create a uniform, accepted definition of AKI; hence RIFLE criteria was born. RIFLE is an acronym of Risk, Injury, Failure, Loss of Kidney Function & End-Stage Kidney Failure.
* In 2004, The Acute Kidney Injury Network (AKIN) was formed. A report of the AKIN proposed the following criteria for AKI.
* The AKIN criteria differ from the RIFLE criteria in several ways. The RIFLE criteria are defined as changes within 7 days, while the AKIN criteria suggest using 48 hours. The AKIN classification includes less severe injury in the criteria and AKIN also avoids using the glomerular filtration rate as a marker in AKI, as there is no dependable way to measure glomerular filtration rate and estimated glomerular filtration rate are unreliable in AKI.
* Haase et al. 2009 in their comparative study between RIFLE and AKIN in cardiac surgery; found no difference between the AKI scores11.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or older who will do prolonged neurosurgical procedure, duration of surgery more than 4 hours and ASA 1-2-3.

Exclusion Criteria:

* refusal of consent, preexisting renal transplantation, preexisting nephrectomy, presence of AKI before neurosurgical procedure, operation less than 4 hours, patients aged under 18 years, pregnancy and ASA 4-5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients aged 18 years or older
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
the occurrence of AKI | 2 days
  BY using AKIN criteria.

REFERENCES:
- [Background] Deng Y, Yuan J, Chi R, Ye H, Zhou D, Wang S, Mai C, Nie Z, Wang L, Zhai Y, Gao L, Zhang D, Hu L, Deng Y, Chen C. The Incidence, Risk Factors and Outcomes of Postoperative Acute Kidney Injury in Neurosurgical Critically Ill Patients. Sci Rep. 2017 Jun 26;7(1):4245. doi: 10.1038/s41598-017-04627-3. PMID 28652590